CLINICAL TRIAL: NCT01679041
Title: A Phase II Study of High Dose Chemotherapy With Autologous Hematopoietic Progenitor Cell Transplant for Multiple Sclerosis That Failed at Least Two Lines of Therapy
Brief Title: High Dose Chemo With Stem Cell Transplant as Treatment for Multiple Sclerosis That Failed Prior Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accruals; PI leaving site
Sponsor: Seah Lim M.D. (Industry)
Responsible Party: Sponsor-Investigator, Seah Lim M.D., Sponsor-Principal Investigator (MD), Texas Oncology Cancer Center
Organization: Texas Oncology Cancer Center (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20112015
Record Dates: First submitted 2012-08-29; First posted 2012-09-05 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Conditioning regimens with Alemtuzumab, Fludarabine, and Cyclophosphamide will be used for all patients.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab 10 mg given IV on day 1 of the 5 day conditional regimen
Drug: Fludarabine — Fludarabine 25mg/m2 daily given IV on days 1-5 of the 5 day conditioning regimen
Drug: Cyclophosphamide — Cyclophosphamide is given 3 gm/m2 for mobilization, and then repeated during 5 day conditioning regimen w/ doses of 50mg/kg/day on days 1-4

SUMMARY:
The purpose of this study is to evaluate the toxicity and the effectiveness of high dose chemotherapy with HPC transplant Multiple Sclerosis that has failed at least two lines of therapy

DETAILED DESCRIPTION:
Multiple sclerosis is an inflammatory autoimmune disease characterized by loss of myelin and axonal damage, having typical contrast-enhanced MRI foci as an imaging counterpart. MS shows three main patterns of clinical course: relapsing/remitting, primary progressive and secondary progressive.Concerning disease pattern, secondary progressive is the standard indication, to avoid overtreatment in relapsing/remitting patients or ineffectual treatment in primary relapsing patients.

Currently, MS is the most common autoimmune disease that have been treated with autologous HPC transplants (Fagius et al, 2009; Burt et al, 2009; Saccardi et al, 2006). More than 350 consecutive cases have been reported by the EBMT over the last decade. Most patients who underwent autologous HPC transplant for MS in the early studies had secondary progressive MS, and relatively fewer had relapsing remitting disease, with a Kurtzke Expanded Disability Status Scale (EDSS) of 3.0-9.5 at the time of transplant. Significant objective and subjective improvements have been reported in up to 70% of these patients.

The following conditioning regimens will be used, with Alemtuzumab, Fludarabine, and Cyclophosphamide will be used for all patients. Prophylaxis of Acyclovir, Levaquin, and Fluconazole will be given to prevent infections. The autologous HPC will be infused within 48-72 hours of completing the chemotherapy. The patients will receive additional supportive care medications and treatments as necessary. Neutrophil engraftment will be defined as the day on which the ANC rises to > 500 cells/ml for two consecutive days. Platelet engraftment will be defined as the first day on which the platelet count rises to > 20,000/ml over a 7-day interval without transfusion support.

ELIGIBILITY:
Inclusion Criteria:

Age between 18-60, inclusive

Patients carry a diagnosis of multiple sclerosis, according to the McDonald's criteria for diagnosis (Polman et al, 2011).

Must have a neurologist providing the primary care for the MS and be willing to be evaluated for the multiple sclerosis by the two neurologists who are the co-investigators in the protocol.

Must be documented to be HIV negative.

An EDSS of 3.5 - 5.5

Patients must be able to give written consent.

Inflammatory disease despite primary disease modifying therapy with at least 6 months of interferon and another disease modifying therapy, including fingolimod,glativamir, natalizumab, and mitoxantrone. Failure is defined as two or more clinical relapses with documented neurologic changes (excluding sensory changes) within the year prior to the study. (NOTE: Relapses must have required treatment with corticosteroids). Failure may also be defined as one relapse (excluding sensory changes) treated with methylprednisone and, on a separate occasion within the previous 12 months, evidence of active inflammation (i.e. gadolinium enhancement on MRI scan of the CNS).

No previous history of allergic reaction to cyclophosphamide, G-CSF or mesna

Patients must not be pregnant

Failure to accept or comprehend irreversible sterility as a potential side effect of therapy.

Life expectancy of more than 6 months

No evidence of myelodysplastic syndrome on peripheral blood smear

Not allergic to cyclophosphamide, mesna, fludarabine or alemtuzumab

Baseline serum creatinine must be <1.5 mg/dL, left ventricular ejection fraction >55%, adequate pulmonary functions (oxygen saturation at room air of >90%), and AST and ALT not > 2x upper limits of normal, and no history of previous or active malignancy, except for localized cutaneous basal or squamous cell carcinoma in situ of the cervix.

Exclusion Criteria:

Diagnosis of primary progressive MS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the toxicity of autologous HPC transplant in patients with multiple sclerosis that have failed at least two lines of disease modifier therapy | At 5 years post transplant
  All follow-up appointments will be carried out at Texas Oncology-Amarillo Cancer Center. Patients will be monitored for clinical toxicities and using laboratory blood tests for renal functions, hepatic functions, and bone marrow functions at At discharge post-transplant, then again at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that 6 monthly until death..

SECONDARY OUTCOMES:
To evaluate the effectiveness of high dose chemotherapy with HPC transplant for multiple sclerosis sclerosis that has failed at least two lines of therapy | Assessed at baseline, tat 3 months, 6 months, 9 months, 12 months, and then after every 12 months until death
  hen rechecked Neurologic evaluations will be carried out in the offices of the two neurology co-Investigators and the information provided to the transplant physicians for record. Patient will also undergo a repeat MRI scan at 3 months, 6 months, 9 months, 12 months, and then after every 12 months until death, after the transplant to evaluate changes in the number of MS plaques. Subsequent MRI scan will be determined by the patient's neurologist as is needed clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Seah Lim, MD, Principal Investigator — Texas Oncology
Locations (3):
- United States (3):
  - Amarillo Diagnostic Clinic, Amarillo, Texas
  - Dr Ruby Saulog, Amarillo, Texas
  - Texas Oncology, Amarillo, Texas

REFERENCES:
- [Background] Burt RK, Loh Y, Cohen B, Stefoski D, Balabanov R, Katsamakis G, Oyama Y, Russell EJ, Stern J, Muraro P, Rose J, Testori A, Bucha J, Jovanovic B, Milanetti F, Storek J, Voltarelli JC, Burns WH. Autologous non-myeloablative haemopoietic stem cell transplantation in relapsing-remitting multiple sclerosis: a phase I/II study. Lancet Neurol. 2009 Mar;8(3):244-53. doi: 10.1016/S1474-4422(09)70017-1. Epub 2009 Jan 29. PMID 19186105
- [Background] Burt RK, Marmont A, Oyama Y, Slavin S, Arnold R, Hiepe F, Fassas A, Snowden J, Schuening F, Myint H, Patel DD, Collier D, Heslop H, Krance R, Statkute L, Verda L, Traynor A, Kozak T, Hintzen RQ, Rose JW, Voltarelli J, Loh Y, Territo M, Cohen BA, Craig RM, Varga J, Barr WG. Randomized controlled trials of autologous hematopoietic stem cell transplantation for autoimmune diseases: the evolution from myeloablative to lymphoablative transplant regimens. Arthritis Rheum. 2006 Dec;54(12):3750-60. doi: 10.1002/art.22256. No abstract available. PMID 17133541
- [Background] Fagius J, Lundgren J, Oberg G. Early highly aggressive MS successfully treated by hematopoietic stem cell transplantation. Mult Scler. 2009 Feb;15(2):229-37. doi: 10.1177/1352458508096875. Epub 2008 Sep 19. PMID 18805841
- [Background] Kimiskidis V, Sakellari I, Tsimourtou V, Kapina V, Papagiannopoulos S, Kazis D, Vlaikidis N, Anagnostopoulos A, Fassas A. Autologous stem-cell transplantation in malignant multiple sclerosis: a case with a favorable long-term outcome. Mult Scler. 2008 Mar;14(2):278-83. doi: 10.1177/1352458507082604. Epub 2007 Oct 17. PMID 17942513
- [Background] Lim SH, Kell J, al-Sabah A, Bashi W, Bailey-Wood R. Peripheral blood stem-cell transplantation for refractory autoimmune thrombocytopenic purpura. Lancet. 1997 Feb 15;349(9050):475. doi: 10.1016/S0140-6736(05)61187-7. No abstract available. PMID 9040585
- [Background] Mancardi GL, Murialdo A, Rossi P, Gualandi F, Martino G, Marmont A, Ciceri F, Schenone A, Parodi RC, Capello E, Comi G, Uccelli A. Autologous stem cell transplantation as rescue therapy in malignant forms of multiple sclerosis. Mult Scler. 2005 Jun;11(3):367-71. doi: 10.1191/1352458505ms1181cr. PMID 15957523
- [Background] Pasquini MC, Griffith LM, Arnold DL, Atkins HL, Bowen JD, Chen JT, Freedman MS, Kraft GH, Mancardi GL, Martin R, Muraro PA, Nash RA, Racke MK, Storek J, Saccardi R. Hematopoietic stem cell transplantation for multiple sclerosis: collaboration of the CIBMTR and EBMT to facilitate international clinical studies. Biol Blood Marrow Transplant. 2010 Aug;16(8):1076-83. doi: 10.1016/j.bbmt.2010.03.012. Epub 2010 Mar 18. PMID 20304084
- [Background] Passweg J, Tyndall A. Autologous stem cell transplantation in autoimmune diseases. Semin Hematol. 2007 Oct;44(4):278-85. doi: 10.1053/j.seminhematol.2007.08.001. PMID 17961728
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Saccardi R, Di Gioia M, Bosi A. Haematopoietic stem cell transplantation for autoimmune disorders. Curr Opin Hematol. 2008 Nov;15(6):594-600. doi: 10.1097/MOH.0b013e3283136700. PMID 18832930
- [Background] Saccardi R, Kozak T, Bocelli-Tyndall C, Fassas A, Kazis A, Havrdova E, Carreras E, Saiz A, Lowenberg B, te Boekhorst PA, Gualandio F, Openshaw H, Longo G, Pagliai F, Massacesi L, Deconink E, Ouyang J, Nagore FJ, Besalduch J, Lisukov IA, Bonini A, Merelli E, Slavino S, Gratwohl A, Passweg J, Tyndall A, Steck AJ, Andolina M, Capobianco M, Martin JL, Lugaresi A, Meucci G, Saez RA, Clark RE, Fernandez MN, Fouillard L, Herstenstein B, Koza V, Cocco E, Baurmann H, Mancardi GL; Autoimmune Diseases Working Party of EBMT. Autologous stem cell transplantation for progressive multiple sclerosis: update of the European Group for Blood and Marrow Transplantation autoimmune diseases working party database. Mult Scler. 2006 Dec;12(6):814-23. doi: 10.1177/1352458506071301. PMID 17263012
- [Background] Tyndall A, Gratwohl A. Adult stem cell transplantation in autoimmune disease. Curr Opin Hematol. 2009 Jul;16(4):285-91. doi: 10.1097/MOH.0b013e32832aacb3. PMID 19465851